CLINICAL TRIAL: NCT01197209
Title: A Phase I Neoadjuvant Study of In-situ REIC/Dkk-3 Therapy Followed By Prostatectomy in Patients With High Risk Localized Prostate Cancer
Brief Title: Neoadjuvant Study of In-situ REIC/Dkk-3 in Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended due to change in development plans and investigator
Sponsor: Momotaro-Gene Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTG-REIC-PC001
Record Dates: First submitted 2010-09-03; First posted 2010-09-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatectomy; Postectomy; Oncology; REIC; Dikkoff; Apoptosis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-REIC/Dkk-3 Arm (Experimental): Active arm on Ad-REIC/Dkk-3
  Interventions: Biological: Ad-REIC/Dkk-3

INTERVENTIONS:
Biological: Ad-REIC/Dkk-3 — REIC (Reduced Expression in Immortalized Cells) protein is down regulated in a variety of cancer cell lines including prostate tumors. The REIC gene is identical to the Dickkopf-3 (Dkk-3) gene that is a member of the Dickkopf gene family. Ad-REIC/Dkk-3 is designed as a viral vector that delivers a DNA plasmid capable of producing intracellular REIC protein. The expression plasmid includes the full-length human cDNA sequence for REIC. The adenovirus vector is a transport mechanism to infuse the REIC/Dkk-3 plasmid into the cell providing a temporary transfusion of REIC protein.

SUMMARY:
This is a phase I neoadjuvant gene therapy followed by prostatectomy, open-label, dose-escalation trial for prostate cancer patients with high risk of local recurrence after radical prostatectomy. Patients entered into this trial will have Prostate Cancer of Clinical stage T1c, T2 or T3 with a Gleason Score of between 7 (4+3) and 10 at the time of enrollment. Patients will receive three 1 mL injections (3 mL total volume) of Ad-REIC/Dkk-3 into the prostate prior to undergoing a radical prostatectomy. Three patients will be treated at each dose level unless a dose-limiting toxicity (DLT) is observed or MFD (defined as 1 x 10e12 vp/treatment) is achieved with expansion for up to 6 more patients at the MTD or MFD.

DETAILED DESCRIPTION:
This is a phase I neoadjuvant gene therapy followed by prostatectomy, open-label, dose-escalation trial for prostate cancer patients with high risk of local recurrence after radical prostatectomy. Patients entered into this trial will have Prostate Cancer of Clinical stage T1c, T2 or T3 with a Gleason Score of between 7 (4+3) and 10 at the time of enrollment.

Patients will receive three 1 mL injections (3 mL total volume) of Ad-REIC/Dkk-3 into the prostate under transrectal ultrasound-guidance (TRUS) and, patients will undergo a radical prostatectomy four weeks after the injection.

Patients will receive treatment at one of three dose levels in a sequential dose-escalating design.

Three patients will be treated at each dose level unless a dose-limiting toxicity (DLT) is observed or MFD (defined as 1 x 10e12 vp/treatment) is achieved. Enrollment will proceed to the next dose level if 0 of 3 patients experiences a DLT; if one of the first 3 patients experiences a DLT, three additional patients will be enrolled until a second patient experiences a DLT (which defines the toxic dose) or until six total patients have been treated at that dose level, whichever comes first. If a second DLT is not experienced within that cohort, dose escalation may continue.

Additional patients will be enrolled a minimum of 14 days after treatment of the first patient in the cohort (sentinel patient).

If 2 DLTs are observed within a cohort, enrollment into the cohort will cease and the dose level immediately preceding that dose will be determined to be the MTD. If 2 non-lethal DLTs are observed in Cohort 1, a lower dose cohort (Cohort -1) may be initiated.

Once the MTD is defined, an additional 3-6 patients may be enrolled at that dose level to further evaluate safety of the MTD.

Patients will undergo a scheduled radical prostatectomy approximately 4 weeks after the Ad-REIC/Dkk-3 injection. The prostate tissue removed will be retained and for those patients treated at the MTD, assessed for REIC expression and evidence of apoptosis by TUNEL staining.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 20 and 75 years (inclusive) with histologically documented clinically localized, adenocarcinoma of the prostate scheduled to undergo a radical prostatectomy.
2. Patient with clinical stage T1c, T2 or T3 with Primary Gleason score of 4 [total Gleason score of between 7 (4+3) and 10] at time of assessment for this trial.
3. Recent (≤ 3 months prior to study entry) negative bone scan and CT scan of abdomen/pelvis.
4. Life expectancy of at least 10 years.
5. In good general health, free from clinically significant illness or disease (as determined by medical/surgical history, physical examination, weight, 12-lead ECG, and clinical laboratory tests)
6. Appropriate surgical candidate for radical prostatectomy and a performance status of ≤ 2 (Zubrod scale)
7. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count ≥ 1,500 and platelet count of ≥ 100,000, adequate hepatic function with a total bilirubin ≤ 1.5 mg/dl and ALT < 4x the upper limits of normal, adequate renal function defined as serum creatinine ≤ 2.0 mg/dl
8. Body Mass Index ≥ 18 and ≤ 35 kg/m2
9. Patients must have normal coagulation profile (PT, PTT) and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants is limited to local use only (for control of central line patency).
10. Patient is willing to refrain from sexual activity or agrees to use a barrier contraceptive device (e.g. condom) after treatment with Ad-REIC/Dkk-3 and until the prostatectomy operation.
11. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the institution.

Exclusion Criteria:

1. Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy or other investigational status drug within the past 4 weeks.
2. Unable to tolerate transrectal ultrasound.
3. Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing causes of death.
4. Patients with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders are not eligible.
5. Patients who are HIV positive or have chronic hepatitis B or C infections are not eligible (because of possible immune effects of these conditions).
6. Patients with a clinical history of primary or secondary immunodeficiency, autoimmune disease or patients taking immunosuppressive drugs such as corticosteroids continuously for > 4 months [> 5 mg hydrocortisone/day] are ineligible. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have a decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. As a result of medical review, physical examination, the Principal Investigator (or medically qualified nominee) considers the subject unfit for the study.

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 7-days
  To define the Maximum Tolerated Dose (MTD) for intertumoral injection (IT) of Ad-REIC/Dkk-3 viral vector.
Safety evaluation of adverse drug experiences compared with historical precedence | 28-days
  To assess the safety of in-situ therapy with REIC/Dkk-3 gene in prostate cancer patients with high risk of local recurrence after radical prostatectomy. Safety events will be evaluated and assessed with regards to causality and in comparison with historical precedence for this patient population.

SECONDARY OUTCOMES:
Pharmacodynamic Efficacy Markers | 28-days
  To assess the effectiveness of Ad-REIC/Dkk-3 in the treatment of prostate cancer as evaluated by the PSA biomarker and histologic examination of extracted prostate tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hall, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- See also: Momotaro-Gene Website — http://www.mt-gene.com